CLINICAL TRIAL: NCT04110470
Title: Definitive Study for Non-inferiority Randomized Control Trial Comparing the Safety and Cost of a Simplified Post-Operative Radiographic (SPOR) Protocol for Selected Fractures
Brief Title: Comparison of the Safety and Cost of a Simplified Post-Operative Radiograph (SPOR) Protocol
Acronym: SPOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS22019 (B2018:067)
Record Dates: First submitted 2018-11-22; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2018-10

CONDITIONS: Fractures, Bone; Fracture Complications; Xray Complication
MeSH Terms: conditions — Fractures, Bone | interventions — X-Rays

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients will receive standard radiographs post-operative day one or two in hospital, as well as radiographs in clinic at two and six weeks.
  Interventions: Diagnostic Test: X-ray
- Treatment Group (Experimental): These patients will not have routine post-operative in hospital radiographs, or radiographs in clinic at two weeks, unless clinically indicated.
  Interventions: Diagnostic Test: No-Xray

INTERVENTIONS:
Diagnostic Test: X-ray — Patients will receive standard radiographs post-operative day one or two in hospital, as well as radiographs in clinic at two and six weeks.
  Arms: Control Group
Diagnostic Test: No-Xray — These patients will not have routine post-operative in hospital radiographs, or radiographs in clinic at two weeks, unless clinically indicated.
  Arms: Treatment Group

SUMMARY:
The standard post-operative radiographic protocol for the monitoring of fractures at Health Sciences Centre includes post-operative in hospital radiographs as well as radiographs at the two week follow up appointment. This is in addition to good quality intra-operative radiographs. With current operative techniques and implants, orthopaedic surgeons can achieve reliably stable internal fixation. In fact, patients are often allowed to take weight through the fractured limb immediately post-operatively. In these cases, redundant post-operative radiographs likely represent an avoidable cost to the system financially, and an avoidable cost to the patient in additional time spent in hospital and unnecessary radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

* At least one lag screw for each fracture line
* At least one compression plate across each fracture line
* Locked intramedullary nail
* Articular/peri-articular fracture with antiglide/under-contoured plate
* Tension band technique (plate included) in simple fracture pattern
* Operating surgeon is confident in fixation construct, despite non-load sharing criteria.

Exclusion Criteria:

* Fracture >21 days old
* Age <18 years, or open growth plates
* Articular fracture with depression
* Multiple orthopaedic fractures
* History or radiographic appearance of osteoporosis/osteopenia or poor operative bone quality
* Likely difficulty with follow-up in first 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1612 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety of a simplified post-operative radiographic protocol for fractures with stable fixation. | At six weeks.
  Incidence of adverse events with a simplified X-ray protocol within the first six weeks of treatment compared to the standard protocol.
  Adverse events are defined as radiographic signs of implant related failure within the first six weeks of treatment and noted on the six week radiographs.
Cost-effectiveness of a simplified post-operative radiographic protocol for fractures with stable fixation. | At six weeks.
  Cost of a simplified X-ray protocol compared to the standard protocol. Cost-effectiveness will be measured by calculating cost of x-ray, patient care and time spent by patients in clinic.

SECONDARY OUTCOMES:
Patient satisfaction: with a simplified post-operative radiographic protocol. | At six weeks.
  A validated 17 question survey tool is used with each question in a 10 centimeter visual analog scale format. Examples of scale ranges (0-10) are provided. The following is a list of some questions asked of participants:
  1. Staff don't seem to listen to anything I tell them during my consultation.
     Agree Disagree
  2. I feel that I'm in good hands when I come to the clinic.
     Agree Disagree
  3. I'm always given a clear explanation of why I am having tests done.
     Agree Disagree
  4. There are some things about my care in the clinic which could be improved.
     Agree Disagree
  5. The person I see in clinic really

CONTACTS AND LOCATIONS:
Overall Officials: Tudor V Tufescu, BSc, MD, FRCSC, Principal Investigator — University of Manitoba

IPD SHARING:
Plan to Share IPD: No